CLINICAL TRIAL: NCT05352321
Title: Multicenter Randomized Controlled Trial of Surgery Plus Target-reduction Chemoradiotherapy vs Regular Chemoradiotherapy for Newly Diagnosed Resectable Nasopharyngeal Carcinoma
Brief Title: Surgery Plus Target-reduction Chemoradiotherapy vs Regular Chemoradiotherapy for Newly Diagnosed Resectable Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Professor, Chief Physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2022-122-01
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Surgery; Target-reduction Chemoradiotherapy; Locally Resectable Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery Plus Target-reduction Chemoradiotherapy (Experimental): Surgery:
  Endoscopic nasopharyngectomy: Radical resection of primary lesion using nasal endoscopy.
  Retropharyngeal lymphadenectomy: Radical retropharyngeal LNs resection using nasal endoscopy or da Vinci robotics.
  Neck lymph node dissection: Selective neck dissection of the region where the positive lymph nodes are located.
  Induction Chemotherapy for stage III-IVa:
  Gemcitabine, 1000 mg/m2, Day 1 and Day 8, Q3W, 3 cycles Cisplatin, 80 mg/m2, Day 1, Q3W, 3 cycles
  Intensity-modulated Radiotherapy with GTV and CTV1 reduction:
  CTV2 : 54.12Gy/33Fr/1.64Gy
  Concurrent Chemotherapy:
  Cisplatin, 100 mg/m2, intravenously, Day 1, Q3W during radiotherapy
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Procedure: surgery; Radiation: Target-reduction intensity-modulated radiotherapy
- Regular Chemoradiotherapy (Active Comparator): Induction Chemotherapy for stage III-IVa:
  Gemcitabine, 1000 mg/m2, intravenously within 30min, Day 1 and Day 8, Q3W, 3 cycles Cisplatin, 80 mg/m2, intravenously, Day 1, Q3W, 3 cycles
  Intensity-modulated Radiotherapy:
  GTVnx (nasopharyngeal lesions): 69.96Gy/33Fr/2.12Gy GTVrnd (retropharyngeal lymph nodes): 69.96Gy/33Fr/2.12Gy GTVnd: 69.96Gy/33Fr/2.12Gy CTV1: 60.60Gy/33Fr/1.82Gy CTV2: 54.12Gy/33Fr/1.64Gy
  Concurrent Chemotherapy:
  Cisplatin, 100 mg/m2, intravenously, Day 1, Q3W during radiotherapy
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Radiation: regular intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Gemcitabine — for induction chemotherapy
Drug: Cisplatin — for induction and concurrent chemotherapy
Radiation: regular intensity-modulated radiotherapy — in active comparator arm
  Arms: Regular Chemoradiotherapy
Procedure: surgery — in experimental arm
  Other Names: Endoscopic nasopharyngectomy; Retropharyngeal lymphadenectomy; Neck lymph node dissection
  Arms: Surgery Plus Target-reduction Chemoradiotherapy
Radiation: Target-reduction intensity-modulated radiotherapy — in experimental arm
  Arms: Surgery Plus Target-reduction Chemoradiotherapy

SUMMARY:
Through a prospective clinical trial, we intend to combine surgery, induction chemotherapy, target-reduction intensity-modulated radiotherapy and concurrent chemotherapy as an experimental treatment for patients with newly diagnosed resectable nasopharyngeal carcinoma to illuminate whether combined surgery could bring patients better local-regional control and lower adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Performance Status Score 0-1 points.
* Non-keratinized carcinoma of the nasopharynx (differentiated or undifferentiated, i.e., WHO type II or III) confirmed histologically and/or cytologically.
* Patients with primary nasopharyngeal lesions evaluated as surgically resectable before chemotherapy, including T1 (tumor limited to nasopharynx), T2 (tumor limited to the surface of parapharyngeal space) and T3 (tumor limited to the bottom wall of sphenoid sinus or pterygoid process). Clinical stage: T1-3N1-3M0, T2-3N0M0 (Stage II-IVA) according to AJCC v8.
* Patients with cervical lymph nodes evaluated as surgically resectable before chemotherapy, including cervical lymph nodes with no invasion (encasement) of the common or ICA, the epidermis, mediastinal structures, prevertebral fascia, or cervical vertebrae.
* Patients with retropharyngeal lymph nodes evaluated as surgically resectable before chemotherapy, including simple RPLNs with intact capsule or RPLNs ≤ 1.5cm with mouth opening range > 4cm.
* Adequate organ function: WBC ≥ 4×10^9 /L, NEUT ≥ 2×10^6 /L, HGB ≥ 9 g/dL, PLT count ≥ 100×10^9/L, TBIL ≤1.5 ULN (TBIL ≤3 ULN for patients with Gilbert Disease), ALT ≤3 ULN, AST ≤3 ULN, ALP ≤3 ULN, ALB ≥ 3 g/dL, INR or APTT≤1.5 ULN, Scr ≤1.5 ULN or Ccr ≥ 60 mL/min.
* Informed Concent signed with willingness to obey the follow-up, treatment, examination and any other programs according to the research protocol.

Exclusion Criteria:

* Diagnosed as recurrent or distant metastatic nasopharyngeal carcinoma or together with any other malignancy.
* Suffering severe cardiopathy or pulmonary dysfunction with cardiac or pulmonary function no more than grade 3.
* Extensive recurrent primary tumour beyond the resectable area such as extensive invasion of the skull base or a distance from the tumour margins to the internal carotid artery of less than 0·5 cm.
* Retropharyngeal lymph node involved or adjacent to primary nasopharyngeal lesions (less than 0·5 cm).
* Unable to cooperate with regular follow-up due to psychological, social, domestic or geological reasons.
* During pregnancy or lactation.
* Other patients that the chief physician considered as illegal for this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Local Regional Relapse-Free Survival (LRRFS) | 3 years
  The LRRFS is evaluated and calculated from the date of random assignment until the day of first local regional relapse or until the date of the last follow-up visit.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Progress-free survival (PFS) | 3 years
  Progress-free survival is calculated from the date of randomization to the date of the first progression of any site or death or censored at the date of the last follow-up.
Distant Metastasis-Free Survival (DMFS) | 3 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Regional Relapse-Free Survival (RRFS) | 3 years
  The RRFS was defined as the duration from the date of random assignment to the date of regional relapse or censored at the date of the last follow-up.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.
Incidence of treatment related acute complications | 1 years
  The proportion of patients with treatment related acute complications according to NCI-CTC5.0 criteria and RTOG criteria.
Incidence of treatment related late complications | 3 years
  The proportion of patients with treatment related late complications according to NCI-CTC5.0 criteria and RTOG criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-yuan Chen, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong